CLINICAL TRIAL: NCT00777335
Title: A Randomized Phase II, Open-label Multicenter Trial of Panobinostat Monotherapy in Women With HER2 Positive Locally Recurrent or Metastatic Breast Cancer
Brief Title: Study of Panobinostat Monotherapy in Women With v-ERB-B2 Avian Erythroblastic Leukemia Viral Oncogene Homolog 2 (HER2) Positive Locally Recurrent or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very low recruitement rate.
Sponsor: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIO 016
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panobinostat i.v. (Experimental)
  Interventions: Drug: Panobinostat - LBH589
- Panobinostat oral (Experimental)
  Interventions: Drug: Panobinostat - LBH589

INTERVENTIONS:
Drug: Panobinostat - LBH589 — Solution for infusion - 25mg/5ml
  Arms: Panobinostat i.v.
Drug: Panobinostat - LBH589 — Hard gelatine capsules - 5mg and 20 mg
  Arms: Panobinostat oral

SUMMARY:
The purpose of the study is to assess the benefit of panobinostat monotherapy given either orally or i.v. to women with HER2-positive locally recurrent or metastatic breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-related procedures
* Women ≥ 18 years old
* Patients with an ECOG performance status of ≤ 2 assessed within 2 weeks prior to randomization
* Histologically or cytologically confirmed invasive breast carcinoma with locally recurrent or radiological evidence of metastatic disease. Locally recurrent disease must not be amenable to resection with curative intent.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) guidelines
* HER2-positive breast cancer patients by local laboratory testing
* Prior trastuzumab-containing regimen (in neoadjuvant and/or adjuvant and/or metastatic settings) regardless of whether trastuzumab was given as monotherapy or in combination with chemotherapy. Any number of prior trastuzumab regimens is acceptable. Additional treatment with lapatinib after or before trastuzumab treatment is permitted, but not mandatory.
* Radiological evidence of relapse or disease progression while on trastuzumab (or lapatinib) or within 12 months of the last dose of adjuvant trastuzumab.
* Complete radiology and tumor assessment within 4 weeks prior to randomization:

  * Chest: Computed Tomography(CT) scan with intravenous contrast if the contrast is not medically contraindicated or Magnetic Resonance Imaging(MRI)
  * Abdomen: CT scan with intravenous and oral contrast if the contrast is not medically contraindicated or MRI
  * Brain: CT scan or MRI
  * Bone: Whole body Bone Scintigraphy
* Up to 2 prior cytotoxic chemotherapy regimens, in addition to neo-adjuvant and adjuvant, for treatment of metastatic or locally recurrent breast cancer (including those cytotoxic chemotherapy treatments in combination with trastuzumab and/or lapatinib)
* Patients must meet the following laboratory criteria within 2 weeks (14 days) prior to randomization:
* Hematology
* Neutrophil count of > 1200/mm3
* Platelet count of > 100,000/mm3
* Hemoglobin ≥ 90 g/L
* Biochemistry
* Aspartate aminotransferase/glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/glutamic pyruvic transaminase(ALT/SGPT) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement
* Serum bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 mL/min
* Serum potassium, sodium, magnesium, phosphorus, total calcium (corrected for serum albumin) or ionized calcium within normal limits for the institution
* Serum albumin ≥ Lower Limit of Normal(LLN) or 30g/L
* Clinically euthyroid function (thyroid-stimulating hormone (TSH) and free T4). (Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism).
* Left Ventricular Ejection Fraction(LVEF) assessment (2-D echocardiogram or Multiple Uptake Gated Acquisition Scan(MUGA) scan) performed within 6 weeks prior to randomization, showing a LVEF value > 50%
* Electrocardiogram performed within 1 week prior to randomization (details about findings on the Electrocardiogram that are not acceptable for participating in the study are reported in the Exclusion criteria section)
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to randomization and agree to appropriate method of pregnancy prevention

Exclusion Criteria:

* Prior Histone Deacetylase(HDAC),Deacetylase(DAC), Heat Shock Protein 90 (HSP90) inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment
* Patients who have received prior chemotherapy or investigational agent within the last 4 weeks prior to randomization (6 weeks for nitrosoureas and mitomycin; 2 weeks for capecitabine)
* Patients who have received prior radiotherapy to ≥ 25% of the bone marrow within the last 4 weeks prior to randomization; local radiotherapy is allowed however all recently irradiated lesions should not be included in the measurable disease assessment
* Patients who have received prior investigational agents within the last 4 weeks prior to randomization
* Patients with unresolved diarrhea ≥CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat
* History of cardiac dysfunction including any one of the following:
* Complete left bundle branch block or necessity for a permanent cardiac pacemaker or congenital long QT syndrome or history or presence of ventricular tachyarrhythmias or clinically significant resting bradycardia (<50 beats per minute) or QTcF > 450 msec on screening electrocardiogram(ECG) or right bundle branch block and left anterior hemiblock (bifascicular block)
* Presence of unstable atrial fibrillation (ventricular response rate >100 bpm). Patients with stable atrial fibrillation are allowed in the study provided they do not meet the other cardiac exclusion criteria
* Previous history angina pectoris or acute myocardial infarction(MI) within 6 months of randomization
* Congestive heart failure (New York Heart Association functional classification III-IV)
* Other clinically significant heart disease (e.g. cardiomyopathy, cardiac artery disease, uncontrolled hypertension, or history of poor compliance with an antihypertensive regimen)
* Acute or chronic liver or renal disease
* Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes mellitus, active untreated or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease including dyspnoea at rest from any cause) that could cause unacceptable safety risks or compromise compliance with the protocol
* Concomitant use of drugs with a risk of causing torsades de pointes where such treatments cannot be discontinued or switched to a different medication prior to starting study drug
* Brain metastases, unless patient randomized on study at least 90 days from completion of brain radiotherapy and / or surgery without radiologic or functional evidence of progressive brain metastases, and off corticosteroids above the dose of 7.5 mg prednisone or equivalent; No concurrent radiotherapy for brain metastasis is allowed
* Clinically significant third space fluid accumulation
* Concurrent bisphosphonates unless if initiated prior to study entry (at least 4 weeks before study randomization)
* Pregnant (i.e., positive beta-human chorionic gonadotropin test) or breast feeding
* Unable to swallow oral medications
* Not willing to use a double barrier method of non-hormonal birth control. Contraception must be used during the study and for 90 days after last dose of study treatment.
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finn, MD, Study Chair — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 28 sites in 4 countries (USA, Canada, France, Belgium).
Period: Overall Study
Arm/Group | Panobinostat Intra-venous (i.v.) | Panobinostat Oral
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panobinostat Intra-venous (i.v.) | Panobinostat Oral | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (20.8) | 59.0 (11.5) | 53.5 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Number; unit: Participants] — 6-point (0 to 5)ordinal scale to assess how the disease affects the daily living abilities of the patient and determine appropriate treatment and prognosis.
  Participants
    PS 0 (Fully active) | 0 | 0 | 0
    PS 1 (Restricted in physically strenuous activity) | 1 | 2 | 3
    PS 2 (Ambulatory and capable of all selfcare) | 1 | 0 | 1
    PS 3 (Capable of only limited selfcare) | 0 | 0 | 0
    PS 4 (Completely disabled) | 0 | 0 | 0
    PS 5 (Dead) | 0 | 0 | 0
Number of lines of prior chemotherapy in metastatic setting [Number; unit: Participants]
  1 line of prior chemotherapy | 0 | 2 | 2
  2 lines of prior chemotherapy | 1 | 0 | 1
  3 lines of prior chemotherapy | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR) Rate (as Determined by the Investigator): the Number of Patients Assigned to a Treatment Arm With a Confirmed Best Response of Complete Response(CR) or Partial Response (PR).
Description: The assessment of OR is based on the response of target lesion, of non-target lesion and on presence of new lesions (RECIST Criteria (V1.0)-assessed by CT scan spiral and bone scan)
  * CR:Disappearance of all target lesions
  * PR:>=30% increase in the sum of the longest diameter (SLD),taking as reference the nadir SLD
  * Progressive Disease (PD):>=20% increase in the SLD, taking as reference the nadir SLD, or the appearance of one or more new lesions
  * Stable Disease(SD):Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the nadir SLD
Time Frame: At screening, every 2 cycles (i.e. 6 weeks) during the first 6 cycles, every 3 cycles (i.e. 9 weeks) during the subsequent cycles and at the End of Treatment (EOT) visit. After the EOT, the tumor assessments should be performed every 9 weeks.
Measure: Number; unit: participants
Arm/Group | Panobinostat Intra-venous (i.v.) | Panobinostat Oral
Number analyzed (Participants) | 2 | 2
participants
  Progressive Disease (PD) | 2 | 1
  Stable Disease (SD) | 0 | 1
  Complete Response (CR) | 0 | 0
  Partial Reponse (PR) | 0 | 0

2. Secondary Outcome: Corrected QT Interval Fridericia's Formula (QTcF)
Description: Prolonged QTcF: QTcF >450 msec and increase of baseline on greater than or equal to 60 msec.
Time Frame: Panobinostat intra-venous (i.v.): All cycles pre-dose measurements. For cycles 1 and 2, post-dose measurements as well. / Panobinostat oral: Pre-dose and post-dose measurements for all cycles. Note: each cycle = 3 weeks
Measure: Number; unit: participants
Arm/Group | Panobinostat Intra-venous (i.v.) | Panobinostat Oral
Number analyzed (Participants) | 2 | 2
participants
  Electrocardiogram QT normal | 1 | 2
  Electrocardiogram QT prolonged | 1 | 0

ADVERSE EVENTS:
Time Frame: The period for collection and reporting of adverse events extends from the time the patient signs the informed consent form (even if the event is not considered to be related to the study drug) until 28 days after the last receipt of the study treatment.
Arm/Group | Panobinostat Intra-venous (i.v.) | Panobinostat Oral
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat Intra-venous (i.v.) (N=2) | Panobinostat Oral (N=2)
Electrocardiogram T wave inversion (Investigations) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat Intra-venous (i.v.) (N=2) | Panobinostat Oral (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 2 (3) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgueusia (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The recruitment rate has shown to be very low worldwide. In total, 4 patients only were recruited, instead of the 132 initially targeted. Due to the very small number of subjects randomized in this study, only descriptive analyses have been made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No